CLINICAL TRIAL: NCT06934135
Title: Randomized, Sham-Controlled Trial of Transcranial Photobiomodulation for Major Depressive Disorder With PET and EEG Biomarker Outcomes.
Brief Title: Trial of Transcranial Photobiomodulation for Depression With PET and EEG Outcomes
Acronym: NITLT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroThera DE (Industry)
Collaborators: Peruvian Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NITLT01
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Depression; Depression, Anxiety; Depressive Disorder; Depressive Disorder, Major
Keywords: Depression, Major Depressive Disorder, Photobiomodulation; FDG-PET, EEG; Near-Infrared Light Therapy, Brain Metabolism; Neurostimulation, Mental Health, Non-Invasive Therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder; Depressive Disorder, Major; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, sham-controlled, parallel-group trial evaluates the effects of transcranial photobiomodulation (tPBM) on depressive symptoms, brain function, and safety in adults with Major Depressive Disorder (MDD). About 112 participants are randomized to one of four arms: high-dose continuous wave (CW, ~350 mW/cm²), low-dose CW (~50 mW/cm²), pulsed wave (PW, peak ~1050 mW/cm²; 42 Hz, 33% duty cycle), or sham. Treatments are delivered 3×/week for 6 weeks (18 sessions) bilaterally over frontal EEG sites AF3/AF4 using 808 nm NIR light (~12 cm² beams).
  The primary outcome is change in HAMD-17 (at baseline, mid, and post-treatment). Secondary outcomes include QIDS-SR16, SDQ, safety metrics, EEG biomarkers (at baseline, mid, and post-treatment), and FDG-PET (baseline and post-treatment) in a 20-participant substudy.
  The study assesses both clinical efficacy and neural mechanisms of action.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, outcome assessors (those evaluating the results), and the sponsor are blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Arm A - Experimental: Continuous Wave (CW, High Dose) (Experimental): Participants receive bilateral tPBM at EEG sites AF3 and AF4 using 808 nm near-infrared light, continuous wave mode. Average irradiance is ~350 mW/cm² (≈4.2 W over two 12 cm² beams). Treatments are delivered twice weekly for 9 weeks (18 sessions total). 429 seconds, 3 times a week for 6 weeks. Delivering to to the brain a total of 3.6 kJ/session, and ~65 kJ/procedure.
  Interventions: Device: Bilateral Near-Infrared Transcranial Photobiomodulation (tPBM)
- Arm B - Experimental: Continuous Wave Low Dose (CW_LOW) (Experimental): Participants receive bilateral tPBM at AF3 and AF4 using 808 nm light in continuous wave mode at reduced average irradiance (~50 mW/cm²; ~1.2 W total). Each 429-second session, three times per week for 6 weeks (18 sessions), delivers ~0.52 kJ/session and ~9.3 kJ total.
  Interventions: Device: Bilateral Near-Infrared Transcranial Photobiomodulation (tPBM)
- Arm C - Experimental: Pulsed Wave (PW) (Experimental): Participants receive bilateral tPBM at AF3 and AF4 using 808 nm light delivered in pulsed mode (42 Hz, 33% duty cycle). Peak irradiance ~1050 mW/cm²; average ~350 mW/cm² (~8.4 W total). Each 429-second session, three times per week for 6 weeks (18 sessions), delivers ~3.6 kJ/session and ~65 kJ total.
  Interventions: Device: Bilateral Near-Infrared Transcranial Photobiomodulation (tPBM)
- Arm D - Sham Comparator: Sham tPBM (Sham Comparator): Participants receive sham stimulation at AF3 and AF4 with an identical-appearing device that emits no therapeutic light. Session length (429 seconds), frequency (3×/week for 6 weeks), and procedures are matched to active arms to maintain blinding.
  Interventions: Device: Bilateral Near-Infrared Transcranial Photobiomodulation (tPBM)

INTERVENTIONS:
Device: Bilateral Near-Infrared Transcranial Photobiomodulation (tPBM) — The system delivers 808 nm near-infrared light via fiber optics through a headset forming ~12 cm² beams at EEG sites AF3/AF4 (dorsolateral prefrontal cortex). Participants are randomized to: (1) Continuous Wave (CW, high dose) ~350 mW/cm² (~8.4 W total); (2) Continuous Wave Low Dose (CW_LOW) ~50 mW/cm² (~1.2 W); (3) Pulsed Wave (PW) peak ~1050 mW/cm², 42 Hz, 33% duty cycle (avg ~350 mW/cm²); or (4) Sham device with identical cues but no light. Sessions last 429 s, 3×/week for 6 weeks (18 total). Sham matches duration/procedures. Outcomes include depressive symptoms (HAMD-17, QIDS, SDQ), FDG-PET, and EEG.
  Other Names: SHAM (Placebo); NIR-TLT

SUMMARY:
Major depressive disorder (MDD) is a leading cause of disability worldwide, and many patients do not achieve adequate benefit from current treatments. Transcranial photobiomodulation (tPBM) is a non-invasive neuromodulation technique that delivers near-infrared (808 nm) light through the scalp to frontal brain regions involved in mood regulation. Preclinical and early clinical studies suggest that tPBM may improve symptoms of depression and enhance cortical function.

This randomized, sham-controlled, parallel-group trial evaluates the efficacy, safety, and neural effects of tPBM in adults with MDD. Participants are assigned to one of four groups: high-dose continuous wave (CW), low-dose continuous wave (CW_LOW), pulsed wave (PW), or sham treatment. Interventions are delivered 3 times a week for 6 weeks (total of 18 sessions) to bilateral frontal scalp sites (AF3 and AF4).

The primary outcome is change in depressive symptoms measured by the Hamilton Depression Rating Scale (HAMD-17) from baseline to week 18. Secondary outcomes include changes in self-reported depression scales (QIDS, SDQ), regional brain glucose metabolism measured by FDG-PET, and resting-state EEG markers. Safety and tolerability are assessed throughout the trial, including adverse events, scalp/site reactions, and suicidality screening.

This study will provide proof-of-concept evidence for the clinical efficacy and mechanistic effects of tPBM in major depression and will inform the design of larger, multicenter clinical trials.

DETAILED DESCRIPTION:
This randomized, sham-controlled, parallel-group clinical trial evaluates the efficacy and safety of transcranial photobiomodulation (tPBM) for adults with major depressive disorder (MDD). Participants are randomly assigned in equal proportions to one of four intervention arms:

1. CW (Continuous Wave, high dose): 808 nm near-infrared laser light delivered continuously at an average irradiance of ~350 mW/cm².
2. CW_LOW (Continuous Wave, low dose): 808 nm laser light delivered continuously at an average irradiance of ~50 mW/cm².
3. PW (Pulsed Wave): 808 nm laser light delivered in pulsed mode at a peak irradiance of ~1050 mW/cm², frequency 42 Hz, with 33% duty cycle.
4. SHAM (Placebo control): Identical headset with no therapeutic light emission, producing only background cues to preserve blinding.

Treatments are administered twice weekly for 9 consecutive weeks (18 sessions total). Each session consists of bilateral application to frontal scalp locations AF3 and AF4 (10-20 EEG system), using circular beams of ~12 cm² per site. The device incorporates standardized positioning and timing protocols to ensure reproducibility across participants.

PET Substudy: A subset of 20 participants undergo 18F-fluorodeoxyglucose positron emission tomography (FDG-PET) imaging at baseline (V0) and post-treatment (V18). Following intravenous tracer injection, participants rest quietly for ~30 minutes prior to scanning. During the uptake and imaging period, participants receive a sequence of 10 minutes of simulated treatment, 10 minutes of their randomized intervention (CW, CW_LOW, PW, or SHAM), and 10 minutes of simulated treatment. The primary PET region of interest is the dorsolateral prefrontal cortex (DLPFC); additional cortical and limbic regions are examined in exploratory analyses.

EEG Assessments: Resting-state electroencephalography (EEG) is recorded at V0, V9, and V18 to evaluate spectral power (delta, theta, alpha, beta bands) and connectivity indices.

Safety Assessments: Safety and tolerability are evaluated at every visit, including collection of adverse events (AEs), serious adverse events (SAEs), scalp/site tolerability ratings (e.g., erythema, discomfort), suicidality screening with the Columbia Suicide Severity Rating Scale (C-SSRS), and reasons for discontinuation.

Hypotheses: The primary hypothesis is that CW tPBM will result in a significantly greater reduction in depressive symptom severity (HAMD-17 total score) compared with SHAM at week 18. Secondary hypotheses include improvement in QIDS and SDQ scores, increased FDG-PET metabolism in DLPFC, and normalization of EEG markers.

ELIGIBILITY:
Inclusion Criteria:

The age of subjects in the study will be between 18 and 75 years (inclusive). Diagnosis of Major Depressive Disorder (MINI). QIDS-C ≥12 at screening. CGI-S ≥4 or higher, i.e., "moderately depressed." Women of childbearing potential must use a double-barrier method of birth control (e.g., condoms plus spermicides) if sexually active.

Written informed consent was obtained from the subject in accordance with local regulations prior to enrollment in this study.

The subject is willing to participate in this study for at least 12 weeks. Subjects must have been on stable doses of antidepressants (if taking any) for at least six weeks before enrollment.

Exclusion Criteria:

A decrease in self-reported SDQ from screening to baseline ≥30%, calculated as [((SDQ_screening-88) - (SDQ_baseline-88)) / (SDQ_screening-88)] ≥30/100. A score of 88 is considered "normal" on the SDQ.

The subject is pregnant or breastfeeding. The subject has failed more than 2 adequate treatments with FDA-approved antidepressants during the current episode according to ATRQ criteria (less than a 50% reduction in depressive symptoms).

Structured psychotherapy focused on treating depression (i.e., CBT or IPT) is allowed if initiated at least 8 weeks before the screening visit.

Substance dependence or abuse in the past 3 months. History of a psychotic disorder or psychotic episode (current psychotic episode as per MINI evaluation).

Bipolar affective disorder (as determined by MINI evaluation). Unstable medical illness, is defined as any medical condition that is not well controlled with standard care medications (e.g., insulin for diabetes mellitus, HCTZ for hypertension).

Active suicidal or homicidal ideation (both intent and plan are present), as determined by C-SSRS screening.

The subject has a significant skin condition (e.g., hemangioma, scleroderma, psoriasis, rash, open wound, or tattoo) on the scalp near any of the procedure sites.

The subject has any type of implant in the head (e.g., stent, clipped aneurysm, embolized AVM, implantable shunt - Hakim valve).

Any use of light-activated medications (photodynamic therapy) within 14 days prior to study enrollment (in the U.S.: Visudyne (verteporfin) - for age-related macular degeneration; Aminolevulinic Acid - for actinic keratosis; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA) - for non-melanoma skin cancer).

Recent history of stroke (within 90 days). The subject had a failed intervention with an FDA-approved device for depression treatment during the current episode (e.g., less than a 50% reduction in depressive symptoms with TMS, ECT, or VNS).

History of dementia, traumatic brain injury (TBI), or any other organic neurological disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Effect on depressive symptoms | Baseline, mid-treatment (Week 3), post-treatment (Week 6), and at 2-week follow-up (Week 8).
  The primary outcome is change in depressive symptom severity in patients with Major Depressive Disorder (MDD), comparing three active doses of near-infrared transcranial light therapy (NIR-TLT) and Sham. Symptoms are measured using the 17-item Hamilton Depression Rating Scale (HAMD-17).

SECONDARY OUTCOMES:
Secondary Outcome Measures | QIDS-SR16 and SDQ: baseline, mid-treatment (Week 3), and post-intervention (Week 6), EEG: baseline, mid-treatment (Week 3), and post-intervention (Week 6), FDG-PET: baseline and post-intervention (Week 6).
  Self-report symptom scales: Quick Inventory of Depressive Symptomatology (QIDS-SR16) and Symptoms of Depression Questionnaire (SDQ), measured at the same intervals.
  Neurophysiological biomarkers:
  Resting-state EEG. Spectral power (delta, theta, alpha, beta) and functional connectivity will be assessed.
  Cerebral glucose metabolism via FDG-PET in a substudy of 20 participants. Primary Region of Interest (ROI): Frontal Lobe. Exploratory ROIs include other cortical/limbic regions.

OTHER OUTCOMES:
Other Pre-Specified Outcomes | Minimally at baseline, mid-treatment (Week 3), and end of treatment (Week 6).
  Composite clinical scores (e.g., Z-score averaging of HAMD-17 and QIDS)
  Safety and tolerability metrics, including:
  Adverse events (AEs) Serious adverse events (SAEs) Scalp/site tolerability (erythema, discomfort) Suicidality assessments using the Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Locations (2):
- Peru (2):
  - Clinica Vesalio, Lima, Lima Province
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima, Lima Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zivin JA, Albers GW, Bornstein N, Chippendale T, Dahlof B, Devlin T, Fisher M, Hacke W, Holt W, Ilic S, Kasner S, Lew R, Nash M, Perez J, Rymer M, Schellinger P, Schneider D, Schwab S, Veltkamp R, Walker M, Streeter J; NeuroThera Effectiveness and Safety Trial-2 Investigators. Effectiveness and safety of transcranial laser therapy for acute ischemic stroke. Stroke. 2009 Apr;40(4):1359-64. doi: 10.1161/STROKEAHA.109.547547. Epub 2009 Feb 20. PMID 19233936
- [Background] Zhang Q, Ma H, Nioka S, Chance B. Study of near infrared technology for intracranial hematoma detection. J Biomed Opt. 2000 Apr;5(2):206-13. doi: 10.1117/1.429988. PMID 10938785
- [Background] Yu W, Naim JO, McGowan M, Ippolito K, Lanzafame RJ. Photomodulation of oxidative metabolism and electron chain enzymes in rat liver mitochondria. Photochem Photobiol. 1997 Dec;66(6):866-71. doi: 10.1111/j.1751-1097.1997.tb03239.x. PMID 9421973
- [Background] Yamaura M, Yao M, Yaroslavsky I, Cohen R, Smotrich M, Kochevar IE. Low level light effects on inflammatory cytokine production by rheumatoid arthritis synoviocytes. Lasers Surg Med. 2009 Apr;41(4):282-90. doi: 10.1002/lsm.20766. PMID 19347944
- [Background] Xu Z, Guo X, Yang Y, Tucker D, Lu Y, Xin N, Zhang G, Yang L, Li J, Du X, Zhang Q, Xu X. Low-Level Laser Irradiation Improves Depression-Like Behaviors in Mice. Mol Neurobiol. 2017 Aug;54(6):4551-4559. doi: 10.1007/s12035-016-9983-2. Epub 2016 Jul 5. PMID 27379735
- [Background] Wu X, Alberico SL, Moges H, De Taboada L, Tedford CE, Anders JJ. Pulsed light irradiation improves behavioral outcome in a rat model of chronic mild stress. Lasers Surg Med. 2012 Mar;44(3):227-32. doi: 10.1002/lsm.22004. Epub 2012 Feb 14. PMID 22334326
- [Background] Thomson, D. J. (1982). Spectrum estimation and harmonic analysis. Proceedings of the IEEE, 70(9), 1055-1096.
- [Background] Simon NM, McNamara K, Chow CW, Maser RS, Papakostas GI, Pollack MH, Nierenberg AA, Fava M, Wong KK. A detailed examination of cytokine abnormalities in Major Depressive Disorder. Eur Neuropsychopharmacol. 2008 Mar;18(3):230-3. doi: 10.1016/j.euroneuro.2007.06.004. Epub 2007 Aug 3. PMID 17681762
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444
- [Background] Shelton RC, Claiborne J, Sidoryk-Wegrzynowicz M, Reddy R, Aschner M, Lewis DA, Mirnics K. Altered expression of genes involved in inflammation and apoptosis in frontal cortex in major depression. Mol Psychiatry. 2011 Jul;16(7):751-62. doi: 10.1038/mp.2010.52. Epub 2010 May 18. PMID 20479761
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Salehpour F, Rasta SH, Mohaddes G, Sadigh-Eteghad S, Salarirad S. Therapeutic effects of 10-HzPulsed wave lasers in rat depression model: A comparison between near-infrared and red wavelengths. Lasers Surg Med. 2016 Sep;48(7):695-705. doi: 10.1002/lsm.22542. Epub 2016 Jul 1. PMID 27367569
- [Background] Salehpour F, Rasta SH. The potential of transcranial photobiomodulation therapy for treatment of major depressive disorder. Rev Neurosci. 2017 May 24;28(4):441-453. doi: 10.1515/revneuro-2016-0087. PMID 28231069
- [Background] Sacher J, Neumann J, Funfstuck T, Soliman A, Villringer A, Schroeter ML. Mapping the depressed brain: a meta-analysis of structural and functional alterations in major depressive disorder. J Affect Disord. 2012 Oct;140(2):142-8. doi: 10.1016/j.jad.2011.08.001. Epub 2011 Sep 3. PMID 21890211
- [Background] Rezin GT, Cardoso MR, Goncalves CL, Scaini G, Fraga DB, Riegel RE, Comim CM, Quevedo J, Streck EL. Inhibition of mitochondrial respiratory chain in brain of rats subjected to an experimental model of depression. Neurochem Int. 2008 Dec;53(6-8):395-400. doi: 10.1016/j.neuint.2008.09.012. Epub 2008 Sep 27. PMID 18940214
- [Background] Ramos-Brieva JA, Cordero Villafafila A. [Validation of the Castillian version of the Hamilton Rating Scale for Depression]. Actas Luso Esp Neurol Psiquiatr Cienc Afines. 1986 Jul-Aug;14(4):324-34. No abstract available. Spanish. PMID 3776732
- [Background] Gili M, Lopez-Navarro E, Homar C, Castro A, Garcia-Toro M, Llobera J, Roca M. Psychometric properties of Spanish version of QIDS-SR16 in depressive patients. Actas Esp Psiquiatr. 2014 Nov-Dec;42(6):292-9. Epub 2014 Nov 1. PMID 25388771
- [Background] Pedrelli P, Blais MA, Alpert JE, Shelton RC, Walker RS, Fava M. Reliability and validity of the Symptoms of Depression Questionnaire (SDQ). CNS Spectr. 2014 Dec;19(6):535-46. doi: 10.1017/S1092852914000406. Epub 2014 Oct 2. PMID 25275853
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858
- [Background] NYU Langone Health (2021, March 5). Transcranial Photobiomodulation for Alzheimer's Disease (TRAP-AD) - Full Text View - ClinicalTrials.gov. Clinical Trials. Retrieved October 22, 2021, from https://clinicaltrials.gov/ct2/show/NCT04784416?term=TRAPAD& draw=2&rank=1
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Morries LD, Cassano P, Henderson TA. Treatments for traumatic brain injury with emphasis on transcranial near-infrared laser phototherapy. Neuropsychiatr Dis Treat. 2015 Aug 20;11:2159-75. doi: 10.2147/NDT.S65809. eCollection 2015. PMID 26347062
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Mohammed HS. Transcranial low-level infrared laser irradiation ameliorates depression induced by reserpine in rats. Lasers Med Sci. 2016 Nov;31(8):1651-1656. doi: 10.1007/s10103-016-2033-5. Epub 2016 Jul 20. PMID 27437987
- [Background] Mochizuki-Oda N, Kataoka Y, Cui Y, Yamada H, Heya M, Awazu K. Effects of near-infra-red laser irradiation on adenosine triphosphate and adenosine diphosphate contents of rat brain tissue. Neurosci Lett. 2002 May 3;323(3):207-10. doi: 10.1016/s0304-3940(02)00159-3. PMID 11959421
- [Background] Michaud CM, McKenna MT, Begg S, Tomijima N, Majmudar M, Bulzacchelli MT, Ebrahim S, Ezzati M, Salomon JA, Kreiser JG, Hogan M, Murray CJ. The burden of disease and injury in the United States 1996. Popul Health Metr. 2006 Oct 18;4:11. doi: 10.1186/1478-7954-4-11. PMID 17049081
- [Background] Lyra V, Parissis J, Kallergi M, Rizos E, Filippatos G, Kremastinos D, Chatziioannou S. 18 F-FDG PET/CT brain glucose metabolism as a marker of different types of depression comorbidity in chronic heart failure patients with impaired systolic function. Eur J Heart Fail. 2020 Nov;22(11):2138-2146. doi: 10.1002/ejhf.1866. Epub 2020 Jun 12. PMID 32530569
- [Background] Lindqvist D, Janelidze S, Hagell P, Erhardt S, Samuelsson M, Minthon L, Hansson O, Bjorkqvist M, Traskman-Bendz L, Brundin L. Interleukin-6 is elevated in the cerebrospinal fluid of suicide attempters and related to symptom severity. Biol Psychiatry. 2009 Aug 1;66(3):287-92. doi: 10.1016/j.biopsych.2009.01.030. Epub 2009 Mar 6. PMID 19268915
- [Background] Levine J, Barak Y, Chengappa KN, Rapoport A, Rebey M, Barak V. Cerebrospinal cytokine levels in patients with acute depression. Neuropsychobiology. 1999 Nov;40(4):171-6. doi: 10.1159/000026615. PMID 10559698
- [Background] Leavitt M, Charles G, Heyman E, Michaels D. HairMax LaserComb laser phototherapy device in the treatment of male androgenetic alopecia: A randomized, double-blind, sham device-controlled, multicentre trial. Clin Drug Investig. 2009;29(5):283-92. doi: 10.2165/00044011-200929050-00001. PMID 19366270
- [Background] Le PN, Ambikairajah E, Epps J, Sethu V, Choi EHC. 2011. Investigation of spectral centroid features for cognitive load classification. Speech Commun. 53:540-551.
- [Background] Kim EA, Kim BG, Yi CH, Kim IG, Chae CH, Kang SK. Macular degeneration in an arc welder. Ind Health. 2007 Apr;45(2):371-3. doi: 10.2486/indhealth.45.371. PMID 17485886
- [Background] Khuman J, Zhang J, Park J, Carroll JD, Donahue C, Whalen MJ. Low-level laser light therapy improves cognitive deficits and inhibits microglial activation after controlled cortical impact in mice. J Neurotrauma. 2012 Jan 20;29(2):408-17. doi: 10.1089/neu.2010.1745. Epub 2011 Sep 21. PMID 21851183
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Iosifescu DV, Bolo NR, Nierenberg AA, Jensen JE, Fava M, Renshaw PF. Brain bioenergetics and response to triiodothyronine augmentation in major depressive disorder. Biol Psychiatry. 2008 Jun 15;63(12):1127-34. doi: 10.1016/j.biopsych.2007.11.020. Epub 2008 Jan 22. PMID 18206856
- [Background] Interian A, Martinez IE, Guarnaccia PJ, Vega WA, Escobar JI. A qualitative analysis of the perception of stigma among Latinos receiving antidepressants. Psychiatr Serv. 2007 Dec;58(12):1591-4. doi: 10.1176/ps.2007.58.12.1591. PMID 18048562
- [Background] Huang ES, Brown SE, Thakur N, Carlisle L, Foley E, Ewigman B, Meltzer DO. Racial/ethnic differences in concerns about current and future medications among patients with type 2 diabetes. Diabetes Care. 2009 Feb;32(2):311-6. doi: 10.2337/dc08-1307. Epub 2008 Nov 18. PMID 19017766
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Hacke W, Schellinger PD, Albers GW, et al. (2014). Transcranial laser therapy in acute stroke
- [Background] Goshen I, Kreisel T, Ben-Menachem-Zidon O, Licht T, Weidenfeld J, Ben-Hur T, Yirmiya R. Brain interleukin-1 mediates chronic stress-induced depression in mice via adrenocortical activation and hippocampal neurogenesis suppression. Mol Psychiatry. 2008 Jul;13(7):717-28. doi: 10.1038/sj.mp.4002055. Epub 2007 Aug 14. PMID 17700577
- [Background] Givens JL, Houston TK, Van Voorhees BW, Ford DE, Cooper LA. Ethnicity and preferences for depression treatment. Gen Hosp Psychiatry. 2007 May-Jun;29(3):182-91. doi: 10.1016/j.genhosppsych.2006.11.002. PMID 17484934
- [Background] Gardner A, Johansson A, Wibom R, Nennesmo I, von Dobeln U, Hagenfeldt L, Hallstrom T. Alterations of mitochondrial function and correlations with personality traits in selected major depressive disorder patients. J Affect Disord. 2003 Sep;76(1-3):55-68. doi: 10.1016/s0165-0327(02)00067-8. PMID 12943934
- [Background] Garcia-Portilla MP, Saiz PA, Bousono M, Bascaran MT, Guzman-Quilo C, Bobes J; en nombre del grupo de validacion de la version espanola de la escala de Funcionamiento Personal y Social (PSP). Validation of the Spanish Personal and Social Performance scale (PSP) in outpatients with stable and unstable schizophrenia. Rev Psiquiatr Salud Ment. 2011 Jan;4(1):9-18. doi: 10.1016/j.rpsm.2010.11.003. Epub 2011 Mar 10. English, Spanish. PMID 23446097
- [Background] Ferrando L, Bobes J, Gibert M, Soto M, Soto O (1998). M.I.N.I. Mini International Neuropsychiatric Interview. Spanish version 5.0.0.DSM-IV. Instituto IAP, Madrid, 1998.
- [Background] Ernesto Roldán-Valadez et al. 18F-FDG PET/CT basics. Definition and normal variants. Gac Méd Méx Vol. 144 No. 2, 2008.
- [Background] De Crescenzo F, Ciliberto M, Menghini D, Treglia G, Ebmeier KP, Janiri L. Is 18F-FDG-PET suitable to predict clinical response to the treatment of geriatric depression? A systematic review of PET studies. Aging Ment Health. 2017 Sep;21(9):889-894. doi: 10.1080/13607863.2016.1247413. Epub 2016 Oct 28. PMID 27792402
- [Background] Desikan RS, Segonne F, Fischl B, Quinn BT, Dickerson BC, Blacker D, Buckner RL, Dale AM, Maguire RP, Hyman BT, Albert MS, Killiany RJ. An automated labeling system for subdividing the human cerebral cortex on MRI scans into gyral based regions of interest. Neuroimage. 2006 Jul 1;31(3):968-80. doi: 10.1016/j.neuroimage.2006.01.021. Epub 2006 Mar 10. PMID 16530430
- [Background] Cummins N, Scherer S, Krajewski J, Schnieder S, Epps J, Quatieri TF (2015). A review of depression and suicide risk assessment using speech analysis. Speech Commun. 71:10-49.
- [Background] Cox RW. AFNI: software for analysis and visualization of functional magnetic resonance neuroimages. Comput Biomed Res. 1996 Jun;29(3):162-73. doi: 10.1006/cbmr.1996.0014. PMID 8812068
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- [Background] Cummins N, Scherer S, Krajewski J, Schnieder S, Epps J, Quatieri TF. (2015). A review of depression and suicide risk assessment using speech analysis. Speech Commun.
- [Background] Cassano P, Petrie SR, Mischoulon D, Cusin C, Katnani H, Yeung A, De Taboada L, Archibald A, Bui E, Baer L, Chang T, Chen J, Pedrelli P, Fisher L, Farabaugh A, Hamblin MR, Alpert JE, Fava M, Iosifescu DV. Transcranial Photobiomodulation for the Treatment of Major Depressive Disorder. The ELATED-2 Pilot Trial. Photomed Laser Surg. 2018 Dec;36(12):634-646. doi: 10.1089/pho.2018.4490. Epub 2018 Oct 20. PMID 30346890
- [Background] Ueng PP, Vincent JR, Kawata EE, Lei CH, Lister RM, Larkins BA. Nucleotide sequence analysis of the genomes of the MAV-PS1 and P-PAV isolates of barley yellow dwarf virus. J Gen Virol. 1992 Feb;73 ( Pt 2):487-92. doi: 10.1099/0022-1317-73-2-487. PMID 1538199
- [Background] Connolly CK, Chan NS. Salbutamol and ipratropium in partially reversible airway obstruction. Br J Dis Chest. 1987 Jan;81(1):55-61. doi: 10.1016/0007-0971(87)90108-2. PMID 2959307
- [Background] Cassano P, Cusin C, Mischoulon D, Hamblin MR, De Taboada L, Pisoni A, Chang T, Yeung A, Ionescu DF, Petrie SR, Nierenberg AA, Fava M, Iosifescu DV. Near-Infrared Transcranial Radiation for Major Depressive Disorder: Proof of Concept Study. Psychiatry J. 2015;2015:352979. doi: 10.1155/2015/352979. Epub 2015 Aug 19. PMID 26356811
- [Background] Caldieraro MA, Sani G, Bui E, Cassano P. Long-Term Near-Infrared Photobiomodulation for Anxious Depression Complicated by Takotsubo Cardiomyopathy. J Clin Psychopharmacol. 2018 Jun;38(3):268-270. doi: 10.1097/JCP.0000000000000883. No abstract available. PMID 29601319
- [Background] Bremner JD, Krystal JH, Putnam FW, Southwick SM, Marmar C, Charney DS, Mazure CM. Measurement of dissociative states with the Clinician-Administered Dissociative States Scale (CADSS). J Trauma Stress. 1998 Jan;11(1):125-36. doi: 10.1023/A:1024465317902. PMID 9479681
- [Background] Araki H, Imaoka A, Kuboyama N, Abiko Y. Reduction of interleukin-6 expression in human synoviocytes and rheumatoid arthritis rat joints by linear polarized near infrared light (Superlizer) irradiation. Laser Ther. 2011;20(4):293-300. doi: 10.5978/islsm.11-or_01. PMID 24155540
- [Background] Allan H. Ropper, Martin A. Samuels, Joshua P. Klein, Sashank Prasad. Adams and Victor. Principles of neurology, Graw-Hill Education, Eleventh edition.
- [Background] Al-Halabí S, Sáiz PA, Burón P, et al. (2016).Validation of the Spanish version of the Columbia-Suicide Severity Rating Scale

DOCUMENTS (2):
  • Study Protocol (2023-12-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT06934135/Prot_000.pdf
  • Informed Consent Form (2023-12-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT06934135/ICF_001.pdf